CLINICAL TRIAL: NCT00963404
Title: Image-guided Tumorboost of Localized Unifocal Bladder Cancer: A Phase I/II Study
Brief Title: Image-Guided Tumorboost of Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRRO IP 070109 DaBlaCa-1; M-20080210
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-01

CONDITIONS: Bladder Neoplasms
Keywords: Image-guided Radiotherapy; Fiducial marker; Adverse effects
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tumor-boost (Experimental): Image-guided tumorboost of the bladder cancer.
  Interventions: Radiation: Radiation boost

INTERVENTIONS:
Radiation: Radiation boost — Radiation boost of the bladder-tumor: 10 Gy/5 fractions, 2 Gy per fraction.

SUMMARY:
The purpose of the study is to increase the radiation dose (Boost) to the bladder tumor. The bladder cancer patients included in the study will undergo tumor demarcation. The bladder demarcations will then be the target for an image-guided boost delivered precisely to the expected tumor site.

ELIGIBILITY:
Inclusion Criteria:

* Muscle invasive bladder cancer (transitional carcinoma)
* Unifocal
* TNM stage T2a-4a, N0-1, M0
* unfit for radical cystectomy

Exclusion Criteria:

* Hyperthyroidism
* Multinodular goiter
* Pregnancy
* Breast feeding
* WHO preformance status more than 2
* Iodine allergy
* MRI or CT contrast media allergy
* Bi-lateral hip-prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Local tumor control | One year

SECONDARY OUTCOMES:
Acute and late adverse effects of the radiotherapy treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jimmi Sondergaard, Principal Investigator — The department of Oncology, Aarhus University Hospital
Locations (4):
- Denmark (4):
  - The department of Oncology, Aarhus University Hospital, Aarhus
  - The department of Oncology, Rigshospitalet, Copenhagen
  - The department of Oncology, Herlev University Hospital, Herlev
  - The department of Oncology, Odense University Hospital, Odense

REFERENCES:
- See also: Related Info — http://www.cirro.dk